CLINICAL TRIAL: NCT05680727
Title: The Role of Individualized Functional Connectivity Targeting in Accelerated Intelligent Neuromodulation Therapy (AINT) for Depression
Brief Title: Individualized Functional Connectivity Targeting in aiTBS for Depression
Acronym: AINT
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Joseph J. Taylor, MD, PhD, Medical Director of TMS, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2022p001650
Record Dates: First submitted 2022-12-13; First posted 2023-01-11 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Depressive Disorder, Major; Depression; Mood Disorders; Mental Disorder; Psychiatric Disorder
Keywords: transcranial magnetic stimulation; accelerated intermittent theta burst stimulation; theta burst stimulation; brain stimulation; neuromodulation; depression; transcranial; TMS; neuronavigation; functional connectivity; neuroimaging
MeSH Terms: conditions — Depressive Disorder, Major; Depression; Mood Disorders; Mental Disorders | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: Parallel-group double-blind randomized controlled trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants will put on a swim cap and undergo treatment site-marking according to standard protocols. All individuals will get two treatment sites marked: 1) Their individualized target based on resting state functional connectivity data, and 2) Beam F3 target based on head measurements. One group will be treated at target #1, and the other group will be treated at target #2.
  Neither group will be able to see the computer screen that shows the neuronavigation in real-time, although they will be able to see their MRI scan on a monitor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- real individualized resting state functional connectivity targeting (Other): Participants in this group will receive aiTBS with neuronavigation to a treatment target identified with individualized resting state functional connectivity.
  Interventions: Procedure: transcranial magnetic stimulation
- sham individualized resting state functional connectivity targeting (Other): Participants in this group will receive aiTBS with neuronavigation to a treatment target identified with head measurements (i.e., Beam F3)
  Interventions: Procedure: transcranial magnetic stimulation

INTERVENTIONS:
Procedure: transcranial magnetic stimulation — Transcranial magnetic stimulation (TMS) is a focal, non-invasive form of brain stimulation that has FDA clearance for depression. In this study, a form of TMS called accelerated intermittent theta burst stimulation will be administered under the supervision of a physician with TMS expertise. This protocol will be modeled after the FDA cleared Stanford Accelerated Intelligent Neuromodulation Therapy (SAINT) protocol, but the patented SAINT rsfc targeting algorithm will not be used for either arm.
  Other Names: TMS; theta burst stimulation; accelerated intermittent theta burst stimulation; aiTBS

SUMMARY:
The goal of this clinical trial is to estimate the importance of neuroimaging in accelerated intermittent theta burst stimulation (aiTBS) for depression. Participants will receive aiTBS treatment, but they will not know if their treatment spot was found with neuroimaging or head measurements.

DETAILED DESCRIPTION:
Techniques for modulating human brain networks are rapidly evolving. One of the most exciting new developments is accelerated intermittent theta burst stimulation (aiTBS), a transcranial magnetic stimulation (TMS) protocol that involves multiple daily treatments rather than gold standard once daily treatment. A specific accelerated iTBS protocol called Stanford Accelerated Intelligent Neuromodulation Therapy (SAINT) was cleared by the FDA in September 2022 based on two pilot studies in which patients with treatment-resistant depression rapidly and robustly improved with SAINT. Many of these patients had been depressed for decades and had not improved with conventional TMS or electroconvulsive therapy. Despite these promising results, two issues may limit SAINT scalability: 1) SAINT has only been tested at a single site in a small number of patients, 2) SAINT has never been tested without individualized resting state functional connectivity (rsfc) targeting, which is not widely available or covered by insurance. In this pilot trial, patients with treatment-resistant depression (n=40) will be randomized to one of two active treatment arms: 1) Real aiTBS with real individualized rsfc targeting, or 2) Real aiTBS with sham individualized rsfc targeting (i.e. conventional TMS targeting based on scalp landmarks). All patients will receive active stimulation, which will facilitate enrollment and reduce ethical concerns about placebo treatment in a vulnerable population when there is existing evidence of treatment efficacy. Patients and clinicians will be blind to group assignment, and blind integrity will be assessed. All patients will undergo MRI scans immediately before treatment and at one month follow up, which aligns with our clinical outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* English proficiency sufficient for informed consent, questionnaires/tasks, and treatment
* Primary diagnosis of major depressive disorder per Diagnostic and Statistical Manual (DSM)-V criteria (MINI International Neuropsychiatric Interview)
* >20 on BDI
* >20 on the MADRS 10, 11
* Moderate to severe level of treatment resistance (Maudsley Staging Method)
* Stable antidepressant medication regimen, or remain medication free, for 4 weeks prior to treatment and to remain on this regimen throughout the study (including all follow-up assessments after the 5-day treatment protocol).
* Primary clinician responsible for psychiatric care before, during, and after the trial
* Agreement to lifestyle considerations
* Abstain from becoming pregnant from screening through end of treatment
* Continue usual intake patterns of caffeine- or xanthine-containing products (e.g., coffee, tea, soft drinks, chocolate) throughout treatment
* Abstain from alcohol for at least 24 hours before the start of each MRI and TMS session
* Abstain from tobacco products during treatment day

Exclusion Criteria:

* Active pregnancy as determined by a urine pregnancy test
* Primary psychiatric diagnosis other than major depressive disorder requiring treatment other than comorbid anxiety disorder
* Those who did not respond to electroconvulsive therapy (ECT) after 8 sessions
* Recent (within 4 weeks) or concurrent use of rapid acting antidepressant agent (ketamine/esketamine/ECT)
* History of:
* Prior exposure to TMS
* Neurosurgical intervention for depression
* Autism spectrum disorder
* Intellectual disability
* Severe cognitive impairment
* Significant neurological illness (e.g., dementia, Parkinson's, Huntington's, brain tumor, seizure disorder, subdural hematoma, multiple sclerosis, brain lesion)
* Untreated or insufficiently treated endocrine disorder
* Treatment with investigational drug or intervention during the study period
* Depth-adjusted TMS treatment dose > 65% maximum stimulator output
* ≥ 30% change in MADRS score between screening and baseline
* Anyone presenting with:
* Mania or hypomania
* Psychosis
* Active suicidal ideation or a suicide attempt (defined by C-SSRS) within the past year
* Neurological lesion
* Contraindications to either TMS or MRI (e.g., metallic implants, severe insomnia > 4 hours per night with hypnotic, etc.).
* Current moderate or severe substance use disorder or demonstrating signs of acute substance withdrawal
* Positive urine drug screen for illicit substances
* Severe borderline personality disorder
* Any other condition deemed by the PI to interfere with the study or increase risk to the participant

Ages: 22 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-07-15 (Actual); Primary Completion 2025-03-17 (Actual); Study Completion 2027-03-17 (Estimated)

PRIMARY OUTCOMES:
Montgomery-Åsberg Depression Rating Scale (MADRS) | one month after treatment
  Depression severity rating scale (0-60, higher numbers indicate higher severity). The primary analysis of the primary outcome will be the effect size (i.e., Cohen's d) of imaging-guided accelerated TMS relative to scalp-targeted TMS. This outcome has not changed since the original grant application for this study. Actual group differences will be explored in a secondary analysis of this primary outcome measure.
  Note added May 2025: The description of the primary outcome measure was clarified. The primary outcome remains unchanged.

SECONDARY OUTCOMES:
Montgomery-Åsberg Depression Rating Scale (MADRS) | immediately after treatment ends
  Depression severity rating scale (0-60, higher numbers indicate higher severity). The primary analysis of the primary outcome will be the effect size of imaging-guided accelerated TMS relative to scalp-targeted TMS. In other words, the "number needed to scan." This outcome has not changed since the original grant application for this study and the data remain blinded at the time of this clarification. Actual group differences will be explored in a secondary analysis of this primary outcome measure.
Beck Depression Inventory (BDI) | immediately after treatment ends and at all subsequent timepoints (1 week, 1 month, 3 months, 6 months, 9 months, 12 months)
  Depression severity rating scales (0-63, higher numbers indicate higher severity)
Quick Inventory of Depressive Symptomatology (QIDS) | immediately after treatment ends and at all subsequent timepoints (1 week, 1 month, 3 months, 6 months, 9 months, 12 months)
  Depression severity rating scales (0-27, higher numbers indicate higher severity)
Change in resting state functional connectivity in the depression network | one month after treatment
  blood oxygen level-dependent (BOLD) signal
Percentage of screened patients from TMS clinical programs who select the accelerated iTBS trial over routine clinical TMS | through study completion, an average of 2 years
  Patient preference measure
Temperament and Character Inventory, Revised 140-item | one month after treatment
  Psychobiologically-based personality inventory which measures seven personality dimensions (harm avoidance, novelty seeking, reward dependence, persistence, self-directedness, cooperativeness, and persistence). For each dimension, this yields a scaled T-score (mean score of 50 with standard deviation of 10). This is an overall estimate of personality traits, and there are no "better" or "worse" traits.
Emotional Conflict Resolution Task | one month after treatment
  Computer task measuring accuracy and reaction time
Learning, Multi-Source Interference Task (MSIT) | one month after treatment
  Computer task measuring accuracy and reaction time
Penn Emotion Recognition Task (ER-40) | one month after treatment
  Computer task measuring accuracy and reaction time
Death Suicide IAT (DSIAT) | one month after treatment
  Computer task measuring reaction time
Beck Anxiety Inventory (BAI) | immediately after treatment ends and at all subsequent timepoints (1 week, 1 month, 3 months, 6 months, 9 months, 12 months)
  Anxiety severity rating scale (0-63, higher numbers indicate higher severity)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph J Taylor, MD, PhD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided
De-identified survey response data and/or neuroimaging data may be shared with collaborators for further analysis.